CLINICAL TRIAL: NCT03419273
Title: Adipose Tissue Inflammation in Individuals Undergoing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Other Study IDs: Bariatric surgery
Record Dates: First submitted 2018-01-20; First posted 2018-02-01 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — We are recruiting only those going through bariatric surgery

SUMMARY:
A growing body of work done over the past few decades has established that adipose tissue as an active endocrine organ which secretes a wide range of metabolic and immunological factors collectively called "adipokines (1)." Importantly, these secreted factors enter into the circulation and have paracrine and autocrine actions, which profoundly impact systemic metabolism (e.g., insulin sensitivity). Additionally, in animals, loss of ovarian hormone production via ovariectomy (similar to menopause in humans) leads to increases in both in adipose tissue mass and in adipose tissue inflammation (2) making this tissue less healthy than that from premenopausal animals. To date, no studies have investigated the effect of menopause on abdominal fat in overweight individuals. Knowing if adipose tissue-specific changes occur with menopause may potentially lead to recommendations or therapeutics to improve women's health post menopause.

DETAILED DESCRIPTION:
Subjects will just have to agree to having a small amount of adipose tissue being removed during the bariatric surgery. The investigators will also collect a blood sample at that time. There will be no other visits for the subject.

ELIGIBILITY:
Inclusion Criteria:

* Women who are premenopausal or who are postmenopausal and have been for at least one year.

Males will be recruited to age match female subjects. All subject are already scheduled to have bariatric surgery at the University of Missouri-Columbia Department of Surgery.

Exclusion Criteria:

* Women who are perimenopausal. Women who are on Hormone Replacement Therapy.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subject are already scheduled to have bariatric surgery at the University of Missouri-Columbia Department of Surgery.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
TNFa | measured in the one sample collected at surgery
  TNFa
Il-6 | measured in the one sample collected at surgery
  Il-6
macrophage | measured in the one sample collected at surgery
  macrophage

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter JW, Barnas JL, Welly R, Spencer N, Pitt J, Vieira-Potter VJ, Kanaley JA. Age, Sex, and Depot-Specific Differences in Adipose-Tissue Estrogen Receptors in Individuals with Obesity. Obesity (Silver Spring). 2020 Sep;28(9):1698-1707. doi: 10.1002/oby.22888. Epub 2020 Jul 31. PMID 32734695